CLINICAL TRIAL: NCT02626819
Title: Improving Weight Management at VA: Enhancing the MOVE!23 for Primary Care (CDA 10-206)
Brief Title: Improving Weight Management at the VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CDP 12-252; CDA 10-206 (Other Grant/Funding Number: Veterans Administration)
Record Dates: First submitted 2015-09-29; First posted 2015-12-10 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: Obesity; Weight Management; Primary Care; Health Coach; iPad; Goal Setting; 5As; technology
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded to intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Receiving MOVE! Toward Your Goals (Experimental): Receiving MOVE! Toward Your Goals intervention (MTG tool, health coaching at baseline, follow-up health coaching calls, potential support of goals from primary care provider)
  Interventions: Behavioral: MOVE! Toward Your Goals
- Arm 2: Receiving Enhanced Usual Care (Active Comparator): Receiving Enhanced Usual Care (standard VA Health Living Messages handouts, potential support of weight management efforts from primary care provider)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: MOVE! Toward Your Goals — Patients will take an online tool accessing weight management and lifestyle behaviors, and will meet with a health coach regularly to establish SMART goals to help them in their weight loss journey. The goals may be supported by the patients' PACT members
  Other Names: MTG arm
  Arms: Arm 1: Receiving MOVE! Toward Your Goals
Behavioral: Enhanced Usual Care — Patients will be given information on "healthy living messages" that were created by the VA, and given more information on specific messages they are interested in from the health coaches, but will not receive official coaching. These messages are the current standard of care at the VA for obesity counseling.
  Other Names: EUC arm
  Arms: Arm 2: Receiving Enhanced Usual Care

SUMMARY:
Compared to the general public, a higher percentage of Veterans are obese or overweight with a weight-related medical condition. The VA currently offers an effective weight management program called MOVE!, but the majority of eligible patients do not attend. Veterans see their primary care providers (PCPs) very frequently, making it an important place to receive information on weight management. However, PCPs often fail to discuss weight management with patients, so interventions are needed to encourage weight management counseling within the team-based care model used in primary care at the VA. Investigators used focus groups, interviews, and other research methods to develop the MOVE! Toward Your Goals (MTG) intervention. This intervention combines online tools, counseling by a health coach, and the team-based care model to deliver weight management information to patients.

Investigators will conduct a randomized controlled trial of 320 Veteran patients and their providers at two VA sites (Manhattan and Brooklyn campuses, New York Harbor Healthcare System) to study the impact of the 12-month MTG intervention when compared to Enhanced Usual Care. Veterans in the MTG intervention arm will take the MTG tool, receive personalized weight management materials, health coach counseling, and go to their scheduled primary care (PC) visit. After the initial visit, MTG-arm Veterans will receive follow up telephone coaching over 12 months. All Veterans will attend follow-up visits at 3, 6 and 12 months to assess body mass index, diet and physical activity, and goal attainment.

The objectives of this study are to: (a) test the impact of the MTG intervention on weight and behavior changes; (b) identify predictors of weight loss in Veterans who use goal setting techniques; and (c) determine the impact of the MTG intervention on primary care team obesity-related counseling practices and attitudes.

DETAILED DESCRIPTION:
Veterans shoulder a disproportionate burden of obesity and its co-morbidities, including diabetes, hypertension, and hyperlipidemia. Modest weight loss in obese patients through diet and exercise improves health and prevents chronic disease, but primary care providers (PCPs) often fail to adequately counsel patients about their weight due to lack of time and training. Thus, tools and brief interventions are needed to support providers' behavior change counseling. The VA currently offers the MOVE! program to treat overweight and obese patients, but only 9% of eligible patients attend. At the same time, Veterans on average see their PCPs 3.6 times per year, which supports the importance of developing primary care (PC)-based interventions. The United States Preventive Services Task force (USPSTF) recommends the use of the 5As framework (Assess, Advise, Agree, Assist, Arrange [5A]) for counseling patients about weight.

Interactive behavior change technologies utilizing expert system software programs are an innovative way to facilitate 5As counseling to promote behavior change in primary care. These programs perform computerized risk, lifestyle, and theory- based, behavioral assessment to provide computer-generated, tailored advice to patients. They also can provide information to healthcare teams.

Collaborative goal setting can be used to achieve behavior change in this intervention. This construct, a critical component of several behavior change theories and models and corresponding to "agree" in the 5As model, has been widely recommended for health promotion in primary care. Investigators did formative work using key informant interviews with several VA Patient Aligned Care Teams (PACT), MOVE! staff, and focus groups with Veterans demonstrated that goal setting is feasible and acceptable to patients and PACT teamlets, and provided insight on barriers to goal setting, and ways to facilitate goal-setting conversations.

During the development phase of this project, investigators developed a primary care-based intervention called MOVE! Toward Your Goals (MTG) to facilitate weight management within primary care and increase adoption of intensive VA programs such as MOVE!. The MTG intervention uses a new MTG software tool (that the investigators developed) delivered on tablets to facilitate 5As-based weight management counseling with a health coach and healthcare team to promote goal-setting, behavior change, and weight loss in the primary care setting. The Veteran also receives follow up with 12 health coaching calls over 1 year.

Investigators will conduct a large, multicenter (Manhattan and Brooklyn campuses, New York Harbor Healthcare System) randomized controlled trial of 320 subjects, who will be randomized to receive either Enhanced Usual Care or the MTG Intervention.

The objectives of this study are to: (a) test the impact of the MTG intervention on weight and behavior changes; (b) identify predictors of weight loss in Veterans who use goal setting techniques; and (c) determine the impact of the MTG intervention on primary care team obesity-related counseling practices and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Has not participated in MOVE! in the past year
* Age 18-69 (this age range represents MOVE! eligibility)
* BMI of 30kg/m2 or a BMI of 25 kg/m2 with obesity-associated condition
* Under the care of PCP with at least 1 prior visit with the provider in the past 12 months
* Access to a telephone
* Able to travel to Brooklyn or Manhattan VA for in-person evaluations at 3, 6, and 12 months

Exclusion Criteria:

* Non-Veterans
* A documented current history of active psychosis or other cognitive issues via International Classification of Diseases (ICD-9) codes
* Diabetes diagnosis via ICD-9 code
* Primary care provider recommends that the patient should not participate
* Severe arthritis, valvular disease, cardiac arrhythmia, pregnancy, and/or other conditions (indicated by PCP) limiting moderate PA
* Self-reported inability to read at a 5th grade level due to literacy level or vision problems

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie R. Jay, MD MS, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (2):
- United States (2):
  - Brooklyn Campus of the VA NY Harbor Healthcare System, Brooklyn, NY, Brooklyn, New York
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jay M, Gutnick D, Squires A, Tagliaferro B, Gerchow L, Savarimuthu S, Chintapalli S, Shedlin MG, Kalet A. In our country tortilla doesn't make us fat: cultural factors influencing lifestyle goal-setting for overweight and obese Urban, Latina patients. J Health Care Poor Underserved. 2014 Nov;25(4):1603-22. doi: 10.1353/hpu.2014.0165. PMID 25418230
- [Background] Levine DM, Savarimuthu S, Squires A, Nicholson J, Jay M. Technology-assisted weight loss interventions in primary care: a systematic review. J Gen Intern Med. 2015 Jan;30(1):107-17. doi: 10.1007/s11606-014-2987-6. Epub 2014 Aug 19. PMID 25134692
- [Background] Acosta A, Azzalin A, Emmons CJ, Shuster JJ, Jay M, Lo MC. Improving residents' clinical approach to obesity: impact of a multidisciplinary didactic curriculum. Postgrad Med J. 2014 Nov;90(1069):630-7. doi: 10.1136/postgradmedj-2014-132821. Epub 2014 Sep 11. PMID 25214540
- [Background] Perez H, Jay MR. Good Midlife Dietary Habits May Increase Likelihood of Healthy Aging - Article Review. Journal of clinical outcomes management : JCOM. 2014 Jan 1; 21(3):105-9.
- [Background] Levine D, Jay MR. Another Win for Veggies - Article Review. Journal of clinical outcomes management : JCOM. 2014 Jan 1; 21(5):207-9.
- [Background] Mateo KF, Jay MR. Access to a Behavioral Weight Loss Website With or Without Group Sessions Increased Weight Loss in Statewide Campaign - Article Review. Journal of clinical outcomes management : JCOM. 2014 Jan 1; 21(8):345-8.
- [Background] Creighton S, Jay MR. Are Non-Nutritive Sweetened Beverages Comparable to Water in Weight Loss Trials. Journal of clinical outcomes management : JCOM. 2014 Jan 1; 21(11):490-2.
- [Background] Jay MR, Chintapalli S, Oi K, Squires A, Sherman S, Kalet A. Identifying barrier and facilitators to improving the implementation of weight management services within a patient-centered medical home. [Abstract]. Journal of general internal medicine. 2014 Apr 25; 29(Supplement 1):S115.
- [Background] Jay MR, Mateo KM, Horne M, Squires A, Kalet A, Sherman S. "In the military, your body and your life aren't your own": Unique factors influencing health behavior change in overweight and obese veterans. Journal of general internal medicine. 2014 Apr 25; 29(Supplement 1):S3.
- [Background] Perez HR, Nick MW, Mateo KM, Sherman S, Kalet A, Jay MR. "None of them apply to me": A usability study of the VA's MOVE!23 online weight management software in Latina Women. Journal of general internal medicine. 2014 Apr 23; 29(Supplement 1):S4.
- [Background] Gerchow L, Tagliaferro B, Squires A, Nicholson J, Savarimuthu SM, Gutnick D, Jay M. Latina food patterns in the United States: a qualitative metasynthesis. Nurs Res. 2014 May-Jun;63(3):182-93. doi: 10.1097/NNR.0000000000000030. PMID 24785246
- [Background] Gutnick D, Reims K, Davis C, Gainforth H, Jay MR, Cole S. Brief Action Planning to Facilitate Behavior Change and Support Patient Self-Management. Journal of clinical outcomes management : JCOM. 2014 Jan 1; 21(1):17-29.
- [Background] Jay M, Chintapalli S, Squires A, Mateo KF, Sherman SE, Kalet AL. Barriers and facilitators to providing primary care-based weight management services in a patient centered medical home for Veterans: a qualitative study. BMC Fam Pract. 2015 Nov 14;16:167. doi: 10.1186/s12875-015-0383-x. PMID 26572125
- [Background] Jay M, Mateo KF, Squires AP, Kalet AL, Sherman SE. Military service and other socioecological factors influencing weight and health behavior change in overweight and obese Veterans: a qualitative study to inform intervention development within primary care at the United States Veterans Health Administration. BMC Obes. 2016 Feb 1;3:5. doi: 10.1186/s40608-016-0087-3. eCollection 2015. PMID 26855786
- [Background] Rogers ES, Sherman SE, Malaspina D, Jay M. Prevalence and Predictors of Obesity-Related Counseling Provided by Outpatient Psychiatrists in the United States. Psychiatr Serv. 2016 Oct 1;67(10):1156-1159. doi: 10.1176/appi.ps.201500345. Epub 2016 Jul 1. PMID 27364811
- [Background] Perez HR, Nick MW, Mateo KF, Squires A, Sherman SE, Kalet A, Jay M. Adapting a weight management tool for Latina women: a usability study of the Veteran Health Administration's MOVE!23 tool. BMC Med Inform Decis Mak. 2016 Oct 5;16(1):128. doi: 10.1186/s12911-016-0368-2. PMID 27716279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Started | 22 | 23
Completed | 18 | 20
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Diagnosed w/ catastrophic illness | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  Participants
    number analyzed (Participants) | 21 | 22 | 43
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 19 | 37
    >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  years
    number analyzed (Participants) | 21 | 22 | 43
    (all) | 53.29 (10.37) | 56.14 (10.73) | 54.74 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  Participants
    number analyzed (Participants) | 21 | 22 | 43
    Female | 5 | 9 | 14
    Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  Participants
    number analyzed (Participants) | 21 | 22 | 43
    Hispanic or Latino | 3 | 6 | 9
    Not Hispanic or Latino | 18 | 15 | 33
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  Participants
    number analyzed (Participants) | 21 | 22 | 43
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 11 | 11 | 22
    White | 4 | 4 | 8
    More than one race | 3 | 6 | 9
    Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: One participant from Arm 2 was removed from the study due to a catastrophic illness, and one participant from Arm 1 officially withdrew from study and did not want data to be used. For these reasons only 43 participants were analyzed.
  kg/m2
    number analyzed (Participants) | 21 | 22 | 43
    (all) | 30.7 (3.4) | 33.0 (5.8) | 31.8 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (kg)
Description: Weight Change from baseline to 3 months. Two weight measurements were taken using a Medline MDR500PHY Physician Digital Scale equipped with height rod. The two weight measurements were averaged. Weight was measured in kilograms and height taken at the baseline, using these two measures Body Mass Index was calculated.
Time Frame: 3 Months
Population: Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputations to adjust for missing data.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 21 | 22
kilograms | -1.06 (1.72) | 0.07 (2.40)
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputation to adjust for missing data

2. Primary Outcome: Weight Change (kg)
Description: Change in weight from baseline to 6-months. Two weight measurements were taken using a Medline MDR500PHY Physician Digital Scale equipped with height rod. The two weight measurements were averaged. Weight was measured in kilograms and height taken at the baseline, using these two measures Body Mass Index was calculated.
Time Frame: 6 Months
Population: Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputation to adjust for missing data
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 21 | 22
kilograms | -1.52 (3.06) | 0.23 (3.64)
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputation to adjust for missing data

3. Primary Outcome: Weight Change (kg)
Description: Change in weight from baseline to the 12-months. Two weight measurements were taken using a Medline MDR500PHY Physician Digital Scale equipped with height rod. The two weight measurements were averaged. Weight was measured in kilograms and height taken at the baseline, using these two measures Body Mass Index was calculated.
Time Frame: 12 months
Population: Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputations to adjust for missing data
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 21 | 22
kilograms | -1.02 (4.16) | 0.74 (4.90)
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Weight change was analyzed using Wilcoxon Rank-Sum test along with multiple imputation to adjust for missing data

4. Primary Outcome: Percent of Patients With Clinically Significant Weight Loss
Description: The percentage of patients who achieve 5-10% weight loss at 3- month study visit.
Time Frame: 3 months
Population: At the 3-months, 6 participants in Arm 1 did not complete the study visits and thus were not included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 15 | 22
Participants | 1 | 2
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Fisher Exact

5. Primary Outcome: Percent of Patients With 2.5% Weight Loss at 6 Months.
Description: Percentage of patients who achieved 2.5% weight loss at 6 months. Weight measured in kg.
Time Frame: 6 months
Population: At the 6-months, 2 participants in Arm 1 and 1 participant in Arm 2 did not complete the study visit and thus were not included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 19 | 21
Participants | 7 | 5
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Fisher Exact

6. Primary Outcome: Percent of Patients With Clinically Significant Weight Loss
Description: The percentage of patients who achieve 5-10% weight loss at 6- month study visit.
Time Frame: 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 19 | 21
Participants | 2 | 1
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Fisher Exact

7. Primary Outcome: Percent of Patients Who Achieved 2.5% Weight Loss
Description: Percentage of patients who achieved 2.5% weight loss at 12 months. Weight measured in kg.
Time Frame: 12 months
Population: At the 12-months, 3 participants in Arm 1 and 2 participants in Arm 2 did not complete the study visit and thus were not included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 18 | 20
Participants | 5 | 4
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Fisher Exact

8. Primary Outcome: Percent of Patients With Clinically Significant Weight Loss
Description: The percentage of patients who achieve 5-10% weight loss at 12- month study visit.
Time Frame: 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
Number analyzed (Participants) | 18 | 20
Participants | 2 | 3
Statistical Analysis 1: Comparison: Arm 1: Receiving MOVE! Toward Your Goals vs Arm 2: Receiving Enhanced Usual Care; Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm 1: Receiving MOVE! Toward Your Goals | Arm 2: Receiving Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

LIMITATIONS AND CAVEATS:
* Small sample size, thus unpowered to see significant results
* Low yield of recruitment
* Research Assistants not blinded to study arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT02626819/Prot_SAP_000.pdf